CLINICAL TRIAL: NCT02985034
Title: Prospective Evaluation of Local Tumor Progression After Radiofrequency Ablation of Hepatocellular Carcinoma: Effectiveness of Immediate Second-Look Evaluation Using Pre-RFA MRI and Post-RFA CT Registration
Brief Title: Safety Margin Assessment After RFA Using the Registration of Pre-ablation MRI and Post-ablation CT
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: SNUH-2010-1412
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: HCC; Liver Tumor
Keywords: HCC; RFA; Liver tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: RFA — Radiofrequency ablation (RFA) is performed according to routine practice, and then safety margin is assessed by a) visual side-by-side comparison between pre-RFA MRI and post-RFA CT, and b) registration software for two modalities.

SUMMARY:
Magnetic resonance imaging (MRI) has been widely used for small liver lesion detection and characterization. In patients who undergo RFA, MRI is often performed before RFA, whereas immediate technical success is usually assessed by CT. Conventional visual assessment of two modalities may be more challenging than being anticipated, because acquisition position, respiration, and spatial resolution differ between the two. Therefore, the study purpose is to evaluate the results of software-assisted ablative margin assessment using registration of different pre-and post-RFA modalities compared with the conventional method of side-by-side MRI-CT comparison in patients with HCCs.

ELIGIBILITY:
Inclusion Criteria:

* patients (≥ 18 years) who were referred to our radiology department for liver tumor RFA
* patients who had liver MR images of sufficient quality for pre-RFA evaluation within 30 days before RFA
* patients with 1-3 tumors (<5 cm)

Exclusion Criteria:

* Child-Pugh class C
* any uncorrected coagulopathy
* hypersensitivity to iodine or other reasons that prevented the performance of post-RFA contrast-enhanced CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver tumor and referred to Radiology for RFA.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Local tumor progression (LTP) | 60 months
  5-year-LTP rate in HCC between sufficient and insufficient ablative margin groups (according to visual assessment and registration software-assisted assessment)

SECONDARY OUTCOMES:
technique efficacy | 1 month after RFA
  Rate of absence of viable tumor on 1-months follow-up CT scan.
immediate technical success on visual assessment | 1 day after RFA
  technical success of RFA on post-RFA CT using side-by-side comparison of pre-RFA MRI and post-RFA CT
immediate technical success on registration-software assessment | 1 day after RFA
  technical success of RFA on post-RFA CT using registration-software assessment between pre-RFA MRI and post-RFA CT

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No